CLINICAL TRIAL: NCT02193074
Title: A Phase 3, Randomized, Double-Blind, Sham-Procedure Controlled Study to Assess the Clinical Efficacy and Safety of ISIS 396443 Administered Intrathecally in Patients With Infantile-onset Spinal Muscular Atrophy
Brief Title: A Study to Assess the Efficacy and Safety of Nusinersen (ISIS 396443) in Infants With Spinal Muscular Atrophy
Acronym: ENDEAR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: After a positive interim analysis, the decision was made to terminate the study early to allow for participants to enroll into an open label study
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 396443-CS3B; 2013-004422-29 (EudraCT Number)
Expanded Access: NCT02865109 (No longer available)
Record Dates: First submitted 2014-07-14; First posted 2014-07-17 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; SMA; SMN; SMNRx; ISIS-SMNRx; ISIS-SMN Rx; ISIS 396443; IONIS-SMNRx; IONIS-SMN Rx; Spinraza; ENDEAR
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nusinersen (Experimental)
  Interventions: Drug: nusinersen
- Sham procedure (Sham Comparator)
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Drug: nusinersen — Administered by intrathecal (IT) injection as specified in the treatment arm.
  Other Names: ISIS 396443; BIIB058; Spinraza; IONIS-SMN Rx; ISIS SMNRx
  Arms: nusinersen
Procedure: Sham procedure — Small needle prick on the lower back at the location where the IT injection is normally made
  Arms: Sham procedure

SUMMARY:
The primary objective of the study is to examine the clinical efficacy of nusinersen (ISIS 396443) administered intrathecally (IT) to participants with infantile-onset with infantile-onset spinal muscular atrophy (SMA). The secondary objective of the study is to examine the safety and tolerability of nusinersen administered intrathecally to participants with infantile-onset SMA.

DETAILED DESCRIPTION:
This study was conducted and the protocol was registered by Ionis Pharmaceuticals, Inc..

In August 2016, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Be born (gestational age) between 37 and 42 weeks
* Be medically diagnosed with spinal muscular atrophy (SMA)
* Have Survival Motor Neuron2 (SMN2) Copy number = 2
* Body weight equal to or greater than 3rd percentile for age using appropriate country-specific guidelines
* Be able to follow all study procedures
* Reside within approximately 9 hours ground-travel distance from a participating study center, for the duration of the study

Key Exclusion Criteria:

* Hypoxemia (oxygen [O2] saturation awake less than 96% or O2 saturation asleep less than 96%, without ventilation support) during screening evaluation
* Clinically significant abnormalities in hematology or clinical chemistry parameters or Electrocardiogram (ECG), as assessed by the Site Investigator, at the Screening visit that would render the participant unsuitable for participation in the study
* Participant's parent or legal guardian is not willing to meet standard of care guidelines (including vaccinations and respiratory syncytial virus prophylaxis if available), nor provide nutritional and respiratory support throughout the study

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Max Age: 210 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2014-08-19 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (31):
- United States (12):
  - UCLA Medical Center, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Hospital, Orlando, Florida
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Duke Children's Hospital, Durham, North Carolina
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia - Neurology, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center/Children's Medical Center Dallas, Dallas, Texas
  - Primary Children's Medical Center (University of Utah), Salt Lake City, Utah
- Australia (2):
  - Sydney Children's Hospital, Sydney, New South Wales
  - Royal Children's Hospital, Children's Neuroscience Centre, Parkville, Victoria
- Hôpital Universitaire des Enfants Reine FABIOLA (HUDERF), Brussels, Belgium
- Canada (2):
  - British Columbia Children's Hospital/UBC, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario
- Institut de Myologie, Paris, France
- Germany (2):
  - Universitatsklinikum Essen, Essen
  - Universtatsklinikum Freiburg, Zentrum fur Kinder-und Jugendmedizin , Abteilung Neuropadiatrie und Muskelerkrankungen, Freiburg im Breisgau
- Italy (2):
  - Istituto Giannina Gaslini, Centro Traslazionale di Miologia e Patologie Neurodegenerative, Genova
  - Pediatric Neurology Unit, Catholic University, Rome
- Japan (2):
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Tokyo Women's Medical University, Tokyo
- Seoul National University Hospital, Seoul, South Korea
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Pediatric Neurology Department, Madrid
- University of Gothenburg, The Queen Silvia Children's Hospital, Gothenburg, Sweden
- Hacettepe Children's Hospital, Ankara, Turkey (Türkiye)
- United Kingdom (2):
  - UCL Institute of Child Health/Great Ormond Street, London
  - MRC Centre for Neuromuscular Diseases at Newcastle, Institute of Genetic Medicine Newcastle University, Newcastle

REFERENCES:
- [Derived] Darras BT, Farrar MA, Mercuri E, Finkel RS, Foster R, Hughes SG, Bhan I, Farwell W, Gheuens S. An Integrated Safety Analysis of Infants and Children with Symptomatic Spinal Muscular Atrophy (SMA) Treated with Nusinersen in Seven Clinical Trials. CNS Drugs. 2019 Sep;33(9):919-932. doi: 10.1007/s40263-019-00656-w. PMID 31420846
- [Derived] Dabbous O, Maru B, Jansen JP, Lorenzi M, Cloutier M, Guerin A, Pivneva I, Wu EQ, Arjunji R, Feltner D, Sproule DM. Survival, Motor Function, and Motor Milestones: Comparison of AVXS-101 Relative to Nusinersen for the Treatment of Infants with Spinal Muscular Atrophy Type 1. Adv Ther. 2019 May;36(5):1164-1176. doi: 10.1007/s12325-019-00923-8. Epub 2019 Mar 16. PMID 30879249
- [Derived] Finkel RS, Mercuri E, Darras BT, Connolly AM, Kuntz NL, Kirschner J, Chiriboga CA, Saito K, Servais L, Tizzano E, Topaloglu H, Tulinius M, Montes J, Glanzman AM, Bishop K, Zhong ZJ, Gheuens S, Bennett CF, Schneider E, Farwell W, De Vivo DC; ENDEAR Study Group. Nusinersen versus Sham Control in Infantile-Onset Spinal Muscular Atrophy. N Engl J Med. 2017 Nov 2;377(18):1723-1732. doi: 10.1056/NEJMoa1702752. PMID 29091570
- [Derived] Finkel RS, Chiriboga CA, Vajsar J, Day JW, Montes J, De Vivo DC, Yamashita M, Rigo F, Hung G, Schneider E, Norris DA, Xia S, Bennett CF, Bishop KM. Treatment of infantile-onset spinal muscular atrophy with nusinersen: a phase 2, open-label, dose-escalation study. Lancet. 2016 Dec 17;388(10063):3017-3026. doi: 10.1016/S0140-6736(16)31408-8. Epub 2016 Dec 7. PMID 27939059
- See also: Cure SMA — http://www.curesma.org
- See also: Muscular Dystrophy Association — http://mda.org/disease/spinal-muscular-atrophy
- See also: National Organization for Rare Diseases — https://www.rarediseases.org
- See also: Clinical Study Report (CSR) Synopsis - a results summary — http://clinicalresearch.biogen.com/Content/Studies/CS3b%20Biogen.com%20Packet.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 149 participants screened, 27 were screening failures. A total of 122 participants enrolled and were randomized; 1 participant withdrew prior to receiving treatment.
Groups:
- Control: Sham procedure administered on Study Days 1, 15, 29, 64, 183, and 302.
- Nusinersen: Nusinersen (2.4 mg/mL) administered as an intrathecal (IT) lumbar puncture injection on Study Days 1, 15, 29, 64, 183, and 302.
Period: Overall Study
Arm/Group | Control | Nusinersen
Started | 41 (Randomized and received double-blind treatment.) | 80 (Randomized and received double-blind treatment.)
Completed During Follow-Up Period | 11 | 26
Completed Due to Early Study Termination | 13 | 39
Completed | 24 | 65
Not Completed | 17 | 15
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 16 | 13

BASELINE CHARACTERISTICS:
Groups:
- Nusinersen: Nusinersen (2.4 mg/mL) administered as an IT lumbar puncture injection on Study Days 1, 15, 29, 64, 183, and 302.
- Total: Total of all reporting groups
Arm/Group | Control | Nusinersen | Total
Number analyzed (Participants) | 41 | 80 | 121
Age, Continuous [Mean (Standard Deviation); unit: days]
  Age at Screening | 164.7 (48.54) | 147.2 (46.85) | 153.1 (47.95)
  Age at First Dose | 180.5 (50.92) | 163.4 (49.57) | 169.2 (50.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 43 | 67
  Male | 17 | 37 | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Motor Milestones Responders
Description: The definition of a motor milestones responder was based on improvement in the motor milestones categories in Section 2 of the Hammersmith Infant Neurological Examination (HINE), with the exclusion of voluntary grasp, as follows:
  (i) subject demonstrates ≥ 2-point increase in the motor milestones category of ability to kick or achievement of maximal score on that category (touching toes), or a 1-point increase in the motor milestones category of head control, rolling, sitting, crawling, standing, or walking, and (ii) among the motor milestone categories, with the exclusion of voluntary grasp, there are more categories where there is improvement as defined in (i) than worsening. (For the category of ability to kick, worsening is defined as ≥ 2-point decrease or decrease to the lowest possible score of no kicking. For the other categories, worsening is defined as ≥ 1-point decrease.) The lowest possible score for the HINE is 0 (zero), and the highest possible score for the HINE is 28.
Time Frame: assessed at the later of the Day 183, Day 302, or Day 394 study visits
Population: Intent-to-treat population: all randomized participants who received ≥ 1 dose of study drug/sham procedure with Day 183, Day 302, or Day 394 data; the last available assessment was used. (Participants who died or withdrew from the study were counted as non-responders and were included in the denominator for the calculation of the percentages.)
Measure: Number; unit: percentage of participants
Arm/Group | Control | Nusinersen
Number analyzed (Participants) | 37 | 73
percentage of participants | 0 | 51
Statistical Analysis 1: Comparison: Control vs Nusinersen; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Difference in percentages = 50.68, 95% CI 2-sided [31.81 to 66.48] — exact unconditional confidence interval

2. Primary Outcome: Time to Death or Permanent Ventilation
Description: Estimated proportion of participants who died or required permanent ventilation by a given study day, based on the Kaplan-Meier product-limit method. Time to death or permanent ventilation was defined as either tracheostomy or ≥ 16 hours ventilation/day continuously for > 21 days in the absence of an acute reversible event. This endpoint was adjudicated by a blinded, independent group of experienced clinicians, the Event Adjudication Committee (EAC), based on review of clinical study data and supporting information. Results are based on all available data.
Time Frame: Day 91, Day 182, Day 273, Day 364, Day 394
Population: Intent-to-treat population: all randomized participants who received ≥ 1 dose of study drug/sham procedure and who died or required permanent ventilation.
Measure: Number; unit: proportion of participants
Arm/Group | Control | Nusinersen
Number analyzed (Participants) | 28 | 31
proportion of participants
  By Day 91 (13 weeks/3 months) | 0.268 | 0.240
  By Day 182 (26 weeks/6 months) | 0.605 | 0.294
  By Day 273 (39 weeks/9 months) | 0.702 | 0.404
  By Day 364 (52 weeks/12 months) | 0.735 | 0.447
  By Day 394 (13 months) | 0.735 | 0.447
Statistical Analysis 1: Comparison: Control vs Nusinersen; Test type: Superiority or Other; p = 0.0046, Log Rank; Based on log-rank test stratified by disease duration
Statistical Analysis 2: Comparison: Control vs Nusinersen; Test type: Superiority or Other; p = 0.0164, Cox proportional hazards model; Based on Cox proportional hazards model adjusted for each subject's disease duration at screening; Hazard Ratio (HR) = 0.530, 95% CI 2-sided [0.3156 to 0.8902]

3. Secondary Outcome: Percentage of Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP-INTEND) Responders
Description: A participants was considered a CHOP-INTEND responder if the change from baseline in CHOP-INTEND total score is ≥ 4 points based on assessment at the later of the Day 183, Day 302, or Day 394 study visits. CHOP-INTEND tests includes 16 items structured to move from easiest to hardest with the grading including gravity eliminated (lower scores) to antigravity movements (higher scores). Total scores range from 0 to 64, with higher scores indicating better movement functioning. Results are based on all available data.
Time Frame: assessed at Baseline and the later of the Day 183, Day 302, or Day 394 study visits
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Control | Nusinersen
Number analyzed (Participants) | 37 | 73
percentage of participants | 3 | 71
Statistical Analysis 1: Comparison: Control vs Nusinersen; Test type: Superiority or Other; p < 0.0001, Fisher Exact; DIfference in percentages = 68.53, 95% CI 2-sided [51.27 to 81.99]

4. Secondary Outcome: Summary of Time to Death
Description: Estimated proportion of participants who died by given duration thresholds, based on the Kaplan-Meier product-limit method.
Time Frame: Day 91, Day 182, Day 273, Day 364, Day 394
Population: Intent-to-treat population: all randomized participants who received ≥ 1 dose of study drug/sham procedure and who died. Results are based on all available data.
Measure: Number; unit: proportion of particiants
Arm/Group | Control | Nusinersen
Number analyzed (Participants) | 16 | 13
proportion of particiants
  by Day 91 | 0.195 | 0.101
  by Day 182 | 0.348 | 0.141
  by Day 273 | 0.382 | 0.173
  by Day 364 | 0.419 | 0.173
  by Day 394 | 0.419 | 0.173
Statistical Analysis 1: Comparison: Control vs Nusinersen; Test type: Superiority or Other; p = 0.0041, Log Rank; Based on log-rank test stratified by disease duration (primary analysis)
Statistical Analysis 2: Comparison: Control vs Nusinersen; Test type: Superiority or Other; p = 0.0082, Cox proportional hazards; Based on Cox proportional hazards model adjusted for each subject's disease duration at screening (sensitivity analysis); Hazard Ratio (HR) = 0.372, 95% CI 2-sided [0.1787 to 0.7745]

5. Secondary Outcome: Percentage of Participants Not Requiring Permanent Ventilation
Time Frame: Up to Day 394
Population: Intent-to-treat population: all randomized participants who received ≥ 1 dose of study drug/sham procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Control | Nusinersen
Number analyzed (Participants) | 41 | 80
percentage of participants | 68 | 77

6. Secondary Outcome: Percentage of Compound Muscular Action Potential (CMAP) Responders
Description: CMAP is an electrophysiological technique that can be used to determine the approximate number of motor neurons in a muscle or group of muscles. A participant was defined as a CMAP responder if the CMAP amplitude at the peroneal nerve was increasing to or maintained at ≥ 1 mV (comparing to the baseline) based on assessment at the later of the Day 183, Day 302, or Day 394 study visits. Results are based on all available data.
Time Frame: assessed at the later of the Day 183, Day 302, or Day 394 study visits
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Control | Nusinersen
Number analyzed (Participants) | 37 | 73
percentage of participants | 5 | 36
Statistical Analysis 1: Comparison: Control vs Nusinersen; Test type: Superiority or Other; p = 0.0004, Fisher Exact; Difference in percentages = 30.21, 95% CI 2-sided [10.35 to 48.09]

7. Secondary Outcome: Time to Death or Permanent Ventilation in the Subgroup of Participants Below the Study Median Disease Duration
Description: Estimated proportion of participants who died or required permanent ventilation (EAC-adjudicated events) among participants below the study median disease duration (13.1 weeks), by given duration thresholds, based on the Kaplan-Meier product-limit method.
Time Frame: Day 91, Day 182, Day 273, Day 364, Day 394
Population: Intent-to-treat population: all randomized participants who received ≥ 1 dose of study drug/sham procedure and were below the study median disease duration.
Measure: Number; unit: proportion of participants
Arm/Group | Control | Nusinersen
Number analyzed (Participants) | 21 | 39
proportion of participants
  by Day 91 | 0.238 | 0.128
  by Day 182 | 0.546 | 0.128
  by Day 273 | 0.697 | 0.228
  by Day 364 | 0.773 | 0.271
  by Day 394 | 0.773 | 0.271
Statistical Analysis 1: Comparison: Control vs Nusinersen; Test type: Superiority or Other; p = 0.0003, Log Rank
Statistical Analysis 2: Comparison: Control vs Nusinersen; Test type: Superiority or Other; p = 0.0014, Cox proportional hazards; Based on Cox proportional hazards model adjusted for each subject's disease duration at screening; Hazard Ratio (HR) = 0.240, 95% CI 2-sided [0.1002 to 0.5753]

8. Secondary Outcome: Time to Death or Permanent Ventilation in the Subgroup of Participants Above the Study Median Disease Duration
Description: Estimated proportion of participants who died or required permanent ventilation (EAC-adjudicated events) among participants above the study median disease duration (13.1 weeks), by given duration thresholds, based on the Kaplan-Meier product-limit method.
Time Frame: Day 91, Day 182, Day 273, Day 364, Day 394
Population: Intent-to-treat population: all randomized participants who received ≥ 1 dose of study drug/sham procedure and were above the study median disease duration.
Measure: Number; unit: proportion of participants
Arm/Group | Control | Nusinersen
Number analyzed (Participants) | 20 | 41
proportion of participants
  by Day 91 | 0.300 | 0.350
  by Day 182 | 0.670 | 0.462
  by Day 273 | 0.725 | 0.584
  by Day 364 | 0.725 | 0.625
  by Day 394 | 0.725 | 0.625
Statistical Analysis 1: Comparison: Control vs Nusinersen; Test type: Superiority or Other; p = 0.3953, Log Rank
Statistical Analysis 2: Comparison: Control vs Nusinersen; Test type: Superiority or Other; p = 0.6268, Cox proportional hazards; Based on Cox proportional hazards model adjusted for each subject's disease duration at screening; Hazard Ratio (HR) = 0.844, 95% CI 2-sided [0.4270 to 1.6698]

9. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs), Serious AEs (SAEs) and Discontinuations Due to AEs
Description: AE: any unfavorable and unintended sign, symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product. SAE: any AE that in the view of either the Investigator or Sponsor, meets any of the following criteria: results in death; is life threatening: that is, poses an immediate risk of death at the time of the event; requires in-patient hospitalization or prolongation of existing hospitalization; results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; results in congenital anomaly or birth defect in the offspring of the participant (whether male or female); is an important medical event in the opinion of the Investigator or Sponsor.
Time Frame: Screening through Day 394 (± 7 days) or early termination
Population: Safety Population: all subjects who received ≥ 1 dose of study drug/sham procedure.
Measure: Number; unit: participants
Arm/Group | Control | Nusinersen
Number analyzed (Participants) | 41 | 80
participants
  Any event | 40 | 77
  Moderate or severe event | 39 | 70
  Severe event | 33 | 45
  Possibly related or related event | 6 | 9
  Related event | 0 | 0
  Serious event | 39 | 61
  Related serious event | 0 | 0
  Treatment discontinuation due to an event | 16 | 13

10. Secondary Outcome: Number of Participants With AEs Corresponding to Changes in Hematology Values
Time Frame: up to Day 394 (± 7 days) or early termination
Population: Safety Population: all subjects who received ≥ 1 dose of study drug/sham procedure.
Measure: Number; unit: participants
Arm/Group | Control | Nusinersen
Number analyzed (Participants) | 41 | 80
participants
  Anemia | 1 | 1
  Neutrophil count increased | 0 | 1
  Leukocytosis | 1 | 0

11. Secondary Outcome: Number of Participants With AEs Corresponding to Changes in Blood Chemistry Values
Time Frame: up to Day 394 (± 7 days) or early termination
Population: Safety Population: all subjects who received ≥ 1 dose of study drug/sham procedure.
Measure: Number; unit: participants
Arm/Group | Control | Nusinersen
Number analyzed (Participants) | 41 | 80
participants
  Blood potassium decreased | 0 | 2
  Liver function test abnormal | 0 | 1
  Alanine aminotransferase increased | 0 | 1
  Aspartate aminotransferase increased | 0 | 1
  Blood chloride decreased | 0 | 1
  Blood iron decreased | 0 | 1
  Blood sodium decreased | 0 | 1
  C-reactive protein increased | 1 | 2
  Hypokalemia | 3 | 2
  Hypoglycemia | 2 | 0
  Hyperglycemia | 1 | 0
  Transaminases increased | 1 | 0

12. Secondary Outcome: Number of Participants Meeting Selected Vital Sign Criteria Post-Baseline
Time Frame: up to Day 394 (± 7 days) or early termination
Population: Safety Population: all subjects who received ≥ 1 dose of study drug/sham procedure and had an assessment.
Measure: Number; unit: participants
Arm/Group | Control | Nusinersen
Number analyzed (Participants) | 41 | 80
participants
  Systolic blood pressure <90 mmHg | 36 | 74
  Systolic blood pressure >140 mmHg | 4 | 4
  Systolic blood pressure >160 mmHg | 0 | 0
  Diastolic blood pressure <50 mmHg | 26 | 71
  Diastolic blood pressure >90 mmHg | 13 | 12
  Diastolic blood pressure >100 mmHg | 3 | 0
  Pulse rate <60 bpm | 0 | 0
  Pulse rate >100 bpm | 41 | 80
  Temperature >38.0 C | 7 | 6
  Temperature <36.0 C | 21 | 45
  Respiratory rate <12 breaths/min | 0 | 0
  Respiratory rate >20 breaths/min | 41 | 80
  Body weight ≥7% decrease from BL | 1 | 4
  Body weight ≥7% increase from BL | 33 | 67

13. Secondary Outcome: Summary of Shifts in 12-lead Electrocardiogram (ECG) Results
Description: Shift to 'abnormal, not clinically significant' includes 'unknown' or 'normal' to 'abnormal, not clinically significant'. Shift to 'abnormal, clinically significant' includes 'unknown' or 'normal' to 'abnormal, clinically significant'.
Time Frame: up to Day 394 (± 7 days) or early termination
Population: Safety Population: all subjects who received ≥ 1 dose of study drug/sham procedure and whose baseline value was not abnormal and who had at least one post-baseline value.
Measure: Number; unit: participants
Arm/Group | Control | Nusinersen
Number analyzed (Participants) | 34 | 65
participants
  Shift to abnormal, not clinically significant | 5 | 17
  Shift to abnormal, clinically significant | 0 | 8
  From unknown to abnormal, clinically significant | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Urinalysis Values
Time Frame: up to Day 394 (± 7 days) or early termination
Population: Safety Population: all subjects who received ≥ 1 dose of study drug/sham procedure.
Measure: Number; unit: participants
Arm/Group | Control | Nusinersen
Number analyzed (Participants) | 41 | 80
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening through Day 394 (± 7 days) or early termination
Description: Treatment-emergent events are presented.
Arm/Group | Control | Nusinersen
Serious Adverse Events (participants affected / at risk) | 39/41 | 61/80
Other Adverse Events (participants affected / at risk) | 35/41 | 70/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=41) | Nusinersen (N=80)
Cardiac arrest (Cardiac disorders) | 2 | 2
Cardio-respiratory arrest (Cardiac disorders) | 5 | 5
Cyanosis (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Death (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 4
Surgical failure (General disorders) | 0 | 1
Bronchiolitis (Infections and infestations) | 1 | 4
Bronchitis (Infections and infestations) | 0 | 4
Bronchitis viral (Infections and infestations) | 0 | 3
Candida sepsis (Infections and infestations) | 1 | 0
Corona virus infection (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 4
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Moraxella infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 19
Pneumonia bacterial (Infections and infestations) | 2 | 3
Pneumonia influenzal (Infections and infestations) | 0 | 1
Pneumonia moraxella (Infections and infestations) | 0 | 1
Pneumonia parainfluenzae viral (Infections and infestations) | 1 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 2 | 6
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 3 | 4
Respiratory tract infection (Infections and infestations) | 1 | 6
Respiratory tract infection viral (Infections and infestations) | 1 | 1
Rhinovirus infection (Infections and infestations) | 2 | 7
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Stoma site abscess (Infections and infestations) | 0 | 1
Systemic infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 0 | 3
Viral infection (Infections and infestations) | 1 | 5
Viral upper respiratory tract infection (Infections and infestations) | 6 | 3
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 0 | 1
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1
Body temperature increased (Investigations) | 1 | 0
Heart rate decreased (Investigations) | 1 | 0
Medical observation (Investigations) | 0 | 2
Oxygen saturation decreased (Investigations) | 2 | 1
Respirovirus test positive (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Feeding disorder of infancy or early childhood (Metabolism and nutrition disorders) | 2 | 2
Feeding intolerance (Metabolism and nutrition disorders) | 0 | 2
Weight gain poor (Metabolism and nutrition disorders) | 2 | 3
Brain injury (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Apnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 | 14
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 8 | 21
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 16 | 20
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=41) | Nusinersen (N=80)
Bradycardia (Cardiac disorders) | 3 | 4
Tachycardia (Cardiac disorders) | 5 | 7
Constipation (Gastrointestinal disorders) | 9 | 28
Diarrhoea (Gastrointestinal disorders) | 7 | 11
Dysphagia (Gastrointestinal disorders) | 9 | 7
Flatulence (Gastrointestinal disorders) | 1 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 10
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 6
Teething (Gastrointestinal disorders) | 3 | 14
Vomiting (Gastrointestinal disorders) | 7 | 11
Oedema (General disorders) | 3 | 0
Pyrexia (General disorders) | 24 | 43
Bacterial tracheitis (Infections and infestations) | 4 | 1
Bronchiolitis (Infections and infestations) | 2 | 4
Candida infection (Infections and infestations) | 3 | 0
Conjunctivitis (Infections and infestations) | 3 | 5
Ear infection (Infections and infestations) | 1 | 5
Influenza (Infections and infestations) | 0 | 5
Nasopharyngitis (Infections and infestations) | 4 | 14
Oral candidiasis (Infections and infestations) | 3 | 7
Pneumonia (Infections and infestations) | 3 | 7
Respiratory tract infection (Infections and infestations) | 2 | 4
Rhinitis (Infections and infestations) | 3 | 2
Rhinovirus infection (Infections and infestations) | 4 | 4
Stoma site infection (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 9 | 22
Urinary tract infection (Infections and infestations) | 0 | 6
Viral infection (Infections and infestations) | 3 | 4
Viral upper respiratory tract infection (Infections and infestations) | 1 | 6
Feeding tube complication (Injury, poisoning and procedural complications) | 3 | 1
Oxygen saturation decreased (Investigations) | 9 | 9
Weight decreased (Investigations) | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 2
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 4 | 6
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.